CLINICAL TRIAL: NCT01307865
Title: Volume Restoration of the Aging Midface With Sculptra Aesthetic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Williams Center Plastic Surgery Specialists (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Edwin F. Williams, III, M.D., Principal Investigator, Williams Center Plastic Surgery Specialists
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFW-001-SA
Record Dates: First submitted 2011-03-02; First posted 2011-03-03 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Problem of Aging
Keywords: midface volume loss; aging of midface; sculptra; sculptra aesthetic; poly-L-lactic acid
MeSH Terms: interventions — New-Fill; poly(lactide)

ARMS (1):
- Sculptra Aesthetic (Experimental): Patients receiving Sculptra Aesthetic
  Interventions: Drug: injectable poly-L-lactic acid

INTERVENTIONS:
Drug: injectable poly-L-lactic acid — Each patient will receive up to 1 vial of Sculptra Aesthetic total to both midface complexes at each of 3 treatment sessions, spaced 6 weeks apart.
  Other Names: Sculptra Aesthetic; Sculptra; Poly-L-lactic acid

SUMMARY:
The purpose of this study is to examine the effect of Sculptra Aesthetic on the cosmetic rejuvenation of the midface complex. The investigators plan to both qualitatively determine the restoration of midface architecture as well as quantitatively document the change in midface volume by employing three-dimensional (3D) surface imaging which critically analyzes volumetric tissue changes. Our hypothesis is that patients who receive Sculptra Aesthetic injections will experience significant improvement in facial midface volume restoration.

* Measure the midfacial volumetric correction from Sculptra Aesthetic treatment, using three-dimensional digital surface imaging
* Determine the mean change from baseline in facial contour via quantitative volumetric measurements
* Correlate volumetric correction with clinical improvement as measured by the Facial Lipoatrophy Panel grading system
* Correlate the mean volumetric change in midfacial treatment area with the amount of product used
* Obtain photographs pre- and post-treatment for the purpose of providing a subject visual aid during the course of treatment
* Collect safety data

ELIGIBILITY:
Inclusion Criteria:

* Age 40-60 years old
* BMI greater than 18.5 and less than 24.9

Exclusion Criteria:

* Age less than 40 years or greater than 60 years
* Prior surgical or non-surgical treatment to the midface within the past 2 years
* Interested in seeking other treatments to the midface during the study period
* Pregnant, lactating, or breast feeding
* Hypersensitivity to poly-L-lactic acid, carboxymethylcellulose, or mannitol
* Allergy to lidocaine or epinephrine
* History of atopy, anaphylaxis, or multiple severe allergies
* Current immunotherapy or history of autoimmune disease
* History of or active stroke or myocardial infarction
* History of or active connective tissue disease
* History of or active bleeding disorders
* History of or active cancer
* Serious abnormalities in laboratory findings
* Active hepatitis
* Active infection or inflammatory process of skin
* History of or risk factors for hypertrophic scarring or keloid formation

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in midfacial volume from Sculptra Aesthetic treatment, using three-dimensional digital surface imaging | 6 mo, 9 mo, 12 mo, 15 mo

SECONDARY OUTCOMES:
Correlate volumetric correction with clinical improvement as measured by the Facial Lipoatrophy Panel grading system | 12 mo
Correlate the mean volumetric change in midfacial volume with the amount of product used | 12 mo
Time course and duration of volumetric correction from Sculptra Aesthetic treatment | 6 mo
Time course and duration of volumetric correction from Sculptra Aesthetic treatment | 9 mo
Time course and duration of volumetric correction from Sculptra Aesthetic treatment | 12 mo
Time course and duration of volumetric correction from Sculptra Aesthetic treatment | 15 mo

CONTACTS AND LOCATIONS:
Overall Officials: Edwin F Williams, MD, Principal Investigator — Williams Center Plastic Surgery Specialists
Locations (1):
- Williams Center Plastic Surgery Specialists, Latham, New York, United States

REFERENCES:
- [Derived] Chen HH, Javadi P, Daines SM, Williams EF 3rd. Quantitative assessment of the longevity of poly-L-lactic acid as a volumizing filler using 3-dimensional photography. JAMA Facial Plast Surg. 2015 Jan-Feb;17(1):39-43. doi: 10.1001/jamafacial.2014.867. PMID 25340593